CLINICAL TRIAL: NCT01160536
Title: The Perceived Impact of Children s Risk Status for Hypertrophic Cardiomyopathy on Families: An Exploratory Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910147; 10-HG-N147
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-08-02

CONDITIONS: Cardiovascular Disease
Keywords: Hypertrophic Cardiomyopathy (HCM); Genetic Testing
MeSH Terms: conditions — Cardiovascular Diseases; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study proposes to describe how children s hypertrophic cardiomyopathy (HCM) risk status affects family functioning, behaviors, and relationships. HCM is the most common inherited cardiovascular single-gene disorder. Individuals with HCM may experience shortness of breath, chest pain, palpitations, dizziness, syncope, heart failure, and arrhythmias predisposing to sudden cardiac death at any age. Notably, HCM is the most common cause of sudden cardiac death in people under 30 years of age. Genetic testing can identify at-risk individuals; however, the impact of potentially life-altering genetic information on families remains largely unexplored. Increasingly, health care providers are providing the testing in children for conditions like HCM that are life-threatening and medically manageable without the benefit of understanding the psychological consequences. The few studies that have been conducted suggest that genetic testing in children may result in changes to family relationships, parental emotional wellbeing, parenting behaviors, and child functioning in a subset of children. One synthesis of these studies suggests that children as a group show little evidence for maladjustment to risk information, but that parents are affected by the carrier status of their children. The proposed study intends to further this body of knowledge by exploring the impact of children s risk status on families with HCM. Health care providers and researchers can inform their work with HCM families by better understanding the potential impact of genetic risk as an important component of families adaptation to the life-threatening information about their children. The families targeted for this exploratory study will be purposively sampled from those that have been aware of the children s risk status or not at-risk status for HCM for at least 3 months. The cross-sectional design is composed of semi-structured interviews with a parent and, separately, with his/her 13 to 23 year-old child who is either a carrier for HCM, a non-carrier, or at 50% risk for being a carrier. The interview will target issues related to the perceived impact of the child s risk status on family functioning, parenting behaviors and relationships. Data from the parent-child dyads will be analyzed for concordance/discordance along parallel themes. The results of this study may facilitate the understanding of the perceived impact of learning children s HCM risk status, which will inform both clinical care and future research. Importantly, since predictive testing in children for adult-onset diseases is generally discouraged, very little is actually known about its impact on families. Therefore, the study of this unique subgroup of an HCM population that uses clinically indicated predictive testing in childhood offers a preliminary opportunity to learn about predictive testing of minors....

DETAILED DESCRIPTION:
This study proposes to describe how children s hypertrophic cardiomyopathy (HCM) risk status affects family functioning, behaviors, and relationships. HCM is the most common inherited cardiovascular single-gene disorder. Individuals with HCM may experience shortness of breath, chest pain, palpitations, dizziness, syncope, heart failure, and arrhythmias predisposing to sudden cardiac death at any age. Notably, HCM is the most common cause of sudden cardiac death in people under 30 years of age. Genetic testing can identify at-risk individuals; however, the impact of potentially life-altering genetic information on families remains largely unexplored. Increasingly, health care providers are providing the testing in children for conditions like HCM that are life-threatening and medically manageable without the benefit of understanding the psychological consequences. The few studies that have been conducted suggest that genetic testing in children may result in changes to family relationships, parental emotional wellbeing, parenting behaviors, and child functioning in a subset of children. One synthesis of these studies suggests that children as a group show little evidence for maladjustment to risk information, but that parents are affected by the carrier status of their children. The proposed study intends to further this body of knowledge by exploring the impact of children s risk status on families with HCM. Health care providers and researchers can inform their work with HCM families by better understanding the potential impact of genetic risk as an important component of families adaptation to the life-threatening information about their children. The families targeted for this exploratory study will be purposively sampled from those that have been aware of the children s risk status or not at-risk status for HCM for at least 3 months. The cross-sectional design is composed of semi-structured interviews with a parent and, separately, with his/her 13 to 23 year-old child who is either a carrier for HCM, a non-carrier, or at 50% risk for being a carrier. The interview will target issues related to the perceived impact of the child s risk status on family functioning, parenting behaviors and relationships. Data from the parent-child dyads will be analyzed for concordance/discordance along parallel themes. The results of this study may facilitate the understanding of the perceived impact of learning children s HCM risk status, which will inform both clinical care and future research. Importantly, since predictive testing in children for adult-onset diseases is generally discouraged, very little is actually known about its impact on families. Therefore, the study of this unique subgroup of an HCM population that uses clinically indicated predictive testing in childhood offers a preliminary opportunity to learn about predictive testing of minors.

ELIGIBILITY:
* INCLUSION CRITERIA:

For Parents:

A parent is eligible to participate in this study if he/she is:

* Biologically related to his/her 13 to 23 year-old child who meets eligibility criteria,
* Self-identified as one of the primary care-takers,
* Aware of the HCM risk status of his/her child(ren) for at least 3 months.
* Cognitive, and
* English-speaking.

For Children:

A child is eligible to participate in this study if he/she is

* Biologically related to his/her eligible parent,
* Between ages 13-23 years old,
* Tested as a minor, and
* Aware of his/her HCM risk status or not at-risk status for at least 3 months,
* Cognitive, and
* English-speaking.

EXCLUSION CRITERIA:

Exclusion criteria: A parent is not eligible to participate in this study if he/she

* Is not biologically related to his/her 13 to 23 year-old child,
* Does not self-identify as one of the primary care-takers,
* Is not aware of the HCM risk status of his/her child(ren) for at least 3 months,
* Is cognitive impaired, or
* Does not speak English.

Exclusion criteria: A child is not eligible to participate I this study if he/she is

* Not biologically related to his/her eligible parent,
* Not between ages 13-to 23 years old,
* Not tested as a minor,
* Not aware of his/her HCM risk status or not at-risk status for at least 3 months,
* Is cognitive impaired, or
* Does not speak English. Note that children who have HCM will not be excluded from the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-06-24; Study Completion 2017-08-02

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- Children's Cardiomyopathy Foundation, Tenafly, New Jersey, United States

REFERENCES:
- [Background] Codori AM, Zawacki KL, Petersen GM, Miglioretti DL, Bacon JA, Trimbath JD, Booker SV, Picarello K, Giardiello FM. Genetic testing for hereditary colorectal cancer in children: long-term psychological effects. Am J Med Genet A. 2003 Jan 15;116A(2):117-28. doi: 10.1002/ajmg.a.10926. PMID 12494429
- [Background] Coffey JS. Parenting a child with chronic illness: a metasynthesis. Pediatr Nurs. 2006 Jan-Feb;32(1):51-9. PMID 16572539
- [Background] Haga SB, Terry SF. Ensuring the safe use of genomic medicine in children. Clin Pediatr (Phila). 2009 Sep;48(7):703-8. doi: 10.1177/0009922809335736. Epub 2009 May 15. PMID 19448129